CLINICAL TRIAL: NCT00005040
Title: Phase II Study of Arsenic Trioxide (NSC #706363) in Relapsed and Refractory Intermediate and High-Grade Non-Hodgkin's Lymphoma
Brief Title: Arsenic Trioxide in Treating Patients With Relapsed or Refractory Non- Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-051; CDR0000067631 (Registry Identifier: PDQ (Physician Data Query)); NCI-T99-0062
Record Dates: First submitted 2000-04-06; First posted 2004-04-12 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma
Keywords: recurrent adult grade III lymphomatoid granulomatosis; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete and partial response rates, duration of complete response, freedom from progression, event free survival, and overall survival in patients with relapsed or refractory intermediate or high grade lymphoma treated with arsenic trioxide. II. Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive arsenic trioxide IV over 2-4 hours for a maximum of 25 cumulative days followed by a rest period of 3-4 weeks. Patients with complete or partial response may receive 6 additional courses in the absence of disease progression or unacceptable toxicity. Patients with minor response (25-50% tumor regression) may also receive further courses of treatment. Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 22-41 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven non-Hodgkin's lymphoma (NHL) that has relapsed following or is resistant to at least 1 standard anticancer therapy or for which no curative therapy exists Intermediate or high grade NHL of one of the following types: Transformed low grade Diffuse small cleaved cell Diffuse large cell (including diffuse mixed cell and immunoblastic large cell) Primary mediastinal B-cell Follicular large cell (follicular center cell or grade III follicular cell) Anaplastic large cell Angiocentric (including nasal T-cell and pulmonary B-cell) Angioimmunoblastic T-cell lymphoma Peripheral T-cell Intestinal T-cell Intravascular lymphomatosis Lymphoblastic Diffuse small noncleaved cell/Burkitt's Adult T-cell leukemia/lymphoma Mantle cell Measurable disease A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 17 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 50 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for at least 4 months after study No active serious infection that is not controlled by antibiotics No grade 3 or worse preexisting neurological abnormality, regardless of causality HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No more than 2 other prior chemotherapy regimens (e.g., one frontline plus one salvage regimen) At least 2 weeks since prior chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 1 month since prior radiotherapy and recovered Surgery: Not specified Other: See Disease Characteristics At least 2 weeks since other prior investigational agents and recovered No concurrent intrathecal drugs

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Straus, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States